CLINICAL TRIAL: NCT06631651
Title: The Effect of Intraoperative Brachioradialis Release on Radiological and Functional Outcomes in Distal Radius Fractures: Long-Term Results
Brief Title: The Effect of Intraoperative Brachioradialis Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hüseyin Emre Tepedelenlioğlu (Other Government)
Responsible Party: Sponsor-Investigator, Hüseyin Emre Tepedelenlioğlu, M.D., Ph.D., Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91610558-604.01.02-
Record Dates: First submitted 2024-06-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Distal Radius Fractures; Brachioradialis Release; Dresdner Scoring
Keywords: Distal Radius Fracture; Brachioralis Release; Wrist Function; DASH Score
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: A retrospective analysis was conducted on 124 patients undergoing surgery for distal radius fractures. Patients were divided into groups based on whether they underwent brachioradialis release during surgery. Pre- and post-operative radiographs were analyzed for anatomical alignment using the Dresdner score. Functional assessments included hand, wrist, and elbow strength, proprioceptive function, and disability levels.
Who Masked: Participant
Masking Description: Patients' ID will/did not be revealed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brachioradialis Release Group (Experimental): During distal radius fracture surgery (open reduction+internal fixation) partial brachioradialis release from the insertion of brachioradialis muscle was performed in order to perform reduction of fracture
  Interventions: Procedure: Brachioradialis release
- Classic (Non-brachioradialis Release) Group (Sham Comparator): During distal radius fracture surgery (open reduction+internal fixation) brachioradialis release was not performed
  Interventions: Procedure: Brachioradialis not released

INTERVENTIONS:
Procedure: Brachioradialis release — During distal radius fracture surgery (open reduction+internal fixation) partial brachioradialis release from the insertion of brachioradialis muscle was performed in order to perform reduction of fracture
  Arms: Brachioradialis Release Group
Procedure: Brachioradialis not released — During distal radius fracture surgery (open reduction+internal fixation) brachioradialis release was not performed.
  Arms: Classic (Non-brachioradialis Release) Group

SUMMARY:
Distal radius fractures are increasingly common, necessitating surgical intervention in many cases for optimal outcomes. Volar plate fixation has emerged as a preferred surgical method due to its effectiveness in promoting faster healing. However, challenges persist in achieving anatomical reduction, particularly concerning the styloid process, where the brachioradialis muscle insertion complicates the procedure. This study explores the impact of intraoperative brachioradialis release on wrist and elbow functions in distal radius fractures.

DETAILED DESCRIPTION:
This two-stage study was conducted in 124 patients who underwent surgery for distal radius fracture between 2011 and 2019. In the first phase, the anatomical alignment of the distal radius was analysed retrospectively. In the second phase, functional assessments of the patients' upper extremities were performed. Patients who underwent open reduction and internal fixation (ARIF) for distal radius end fractures and who agreed to participate in the study were included. Patients who were treated with a method other than ARIF, who had bilateral injuries (valid only for the second phase), who had a fracture in a bone other than the radius, and who had any other neurological or orthopaedic disorder that would affect the assessment were not included in the study.

For the first phase, 124 patients were divided into 2 groups: patients with brachioradialis release (76 patients) and patients without brachioradialis release (38 patients). The release of the brachioradialis muscle was achieved through partial release from its insertion into the styloid process, rather than through Z-plasty. In both groups, the pre- and post-operative radiographs of the operated patients were analysed and the operative times of the operations were recorded. The Dresdner score was calculated by measuring the preoperative and postoperative joint grading, radial tilt angle, palmar tilt angle and ulnar variance on the radiographs. A lower Dresdner score indicated better anatomical alignment.

For the second phase, 124 patients were contacted by telephone. Sixty-one patients who could not be reached or did not meet the inclusion criteria were excluded from the study. The remaining 63 patients were divided into two groups: brachioradialis release and non-brachioradialis release.

In the second stage, hand, wrist and elbow strength, proprioceptive function and disability level of the patients were assessed as functional assessments. The Jebsen Hand Function Test (JEFT) was used to assess hand function.

Wrist flexion-extension, elbow flexion-extension and forearm supination-pronation forces were assessed using an isokinetic dynamometer (Cybex NORM®; Humac, CA, Computer Sports Medicine, Inc., Stoughton, MA).

Elbow flexion-extension strength measurements were conducted while the patient was lying supine on the platform of the isokinetic dynamometer.

Forearm supination-pronation force measurement was performed using an isokinetic dynamometer.

Functional forces of the hand, including key pinch, palmar pinch, tip pinch, and gross grip forces, were evaluated.

Wrist proprioception was assessed by measuring active joint position sense (AJPS).

To evaluate the participants' disability during daily activities, the Turkish version of the Disability Assessment of Arm, Shoulder and Hand Injury Questionnaire (DASH-T) was used.

Statistical Analysis

SPSS 22.0 statistical package was used for the statistical analysis of the data. The normal distribution of the data was assessed using histogram plots, normal Q-Q plots with correction, coefficients of skewness and kurtosis, coefficient of variance and the Shapiro-Wilk test. In the descriptive section of the statistical analysis of the data, categorical variables were presented with numbers, continuous variables with mean and standard deviation for normally distributed variables, and median (minimum-maximum) for non-normally distributed variables. For comparisons between groups, parametric and non-parametric data, the independent samples t-test and the Mann-Whitney U test were used. Changes in parametric variables with repeated measurements were compared between groups using an ordered samples t-test. In this study, the statistical significance level was accepted as p<0.05 with 95% confidence interval. The effect size was expressed as the (eta2) value.

ELIGIBILITY:
Inclusion Criteria:

Voluntary patients with distal radius fractures requiring operation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Operation time | 9 months
  To compare the time taken by the surgical methods, the operation times were compared. For this, the start and end times of the operation were analyzed
Anatomical alignment | 9 months
  Dresdner score was calculated by measuring preoperative and postoperative joint grading, radial inclination angle, palmar inclination angle and ulnar variance on radiography.
Strength Tests | 9 months
  Hand, wrist, forearm, and elbow strengths were evaluated with iskoniteic dynamometer
Proprioception measurement | 9 months
  Hand, wrist, forearm, and elbow proprioceptions were evaluated with iskoniteic dynamometer
functional capacity | 9 months
  Jebsen hand function test was performed to evaluate hand function.
Disability level | 9 months
  The Turkish version of the Disability Assessment of Arm, Shoulder and Hand Injury Questionnaire (DASH-T) was used to assess the participants' disability during activities of daily living.
pinch and grip forces | 9 months
  Key pinch, palmar pinch, tip pinch and gross grip strengths were evaluated with a dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik Şehir Hastanesi, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hagenaars T, Van Oijen GW, Roerdink WH, Vegt PA, Vroemen JP, Verhofstad MH, Van Lieshout EM. Functional recovery after treatment of extra-articular distal radius fractures in the elderly using the IlluminOss(R) System (IO-Wrist); a multicenter prospective observational study. BMC Musculoskelet Disord. 2016 May 27;17:235. doi: 10.1186/s12891-016-1077-9. PMID 27233355
- [Result] Walenkamp MM, Vos LM, Strackee SD, Goslings JC, Schep NW. The Unstable Distal Radius Fracture-How Do We Define It? A Systematic Review. J Wrist Surg. 2015 Nov;4(4):307-16. doi: 10.1055/s-0035-1556860. PMID 26649263
- [Result] Zhou J, Tang W, Li D, Wu Y. Morphological characteristics of different types of distal radius die-punch fractures based on three-column theory. J Orthop Surg Res. 2019 Nov 27;14(1):390. doi: 10.1186/s13018-019-1453-x. PMID 31775810
- [Result] Park MJ, Cooney WP 3rd, Hahn ME, Looi KP, An KN. The effects of dorsally angulated distal radius fractures on carpal kinematics. J Hand Surg Am. 2002 Mar;27(2):223-32. doi: 10.1053/jhsu.2002.32083. PMID 11901381
- [Result] Quinn SF, Murray W, Watkins T, Kloss J. CT for determining the results of treatment of fractures of the wrist. AJR Am J Roentgenol. 1987 Jul;149(1):109-11. doi: 10.2214/ajr.149.1.109. PMID 3495968
- [Result] Fok MW, Klausmeyer MA, Fernandez DL, Orbay JL, Bergada AL. Volar plate fixation of intra-articular distal radius fractures: a retrospective study. J Wrist Surg. 2013 Aug;2(3):247-54. doi: 10.1055/s-0033-1350086. PMID 24436824
- [Result] Kumar S, Khan AN, Sonanis SV. Radiographic and functional evaluation of low profile dorsal versus volar plating for distal radius fractures. J Orthop. 2016 Jul 19;13(4):376-82. doi: 10.1016/j.jor.2016.06.017. eCollection 2016 Dec. PMID 27504057
- [Result] Roh YH, Lee BK, Baek JR, Noh JH, Gong HS, Baek GH. A randomized comparison of volar plate and external fixation for intra-articular distal radius fractures. J Hand Surg Am. 2015 Jan;40(1):34-41. doi: 10.1016/j.jhsa.2014.09.025. Epub 2014 Oct 29. PMID 25446409
- [Result] Chan YH, Foo TL, Yeo CJ, Chew WY. Comparison between cast immobilization versus volar locking plate fixation of distal radius fractures in active elderly patients, the Asian perspective. Hand Surg. 2014;19(1):19-23. doi: 10.1142/S021881041450004X. PMID 24641736
- [Result] Protopsaltis TS, Ruch DS. Volar approach to distal radius fractures. J Hand Surg Am. 2008 Jul-Aug;33(6):958-65. doi: 10.1016/j.jhsa.2008.04.018. PMID 18656773
- [Result] Koh S, Andersen CR, Buford WL Jr, Patterson RM, Viegas SF. Anatomy of the distal brachioradialis and its potential relationship to distal radius fracture. J Hand Surg Am. 2006 Jan;31(1):2-8. doi: 10.1016/j.jhsa.2005.08.012. PMID 16443096
- [Result] Sarmiento A. The brachioradialis as a deforming force in Colles' fractures. Clin Orthop Relat Res. 1965 Jan-Feb;38:86-92. No abstract available. PMID 5889097
- [Result] Orbay JL, Fernandez DL. Volar fixation for dorsally displaced fractures of the distal radius: a preliminary report. J Hand Surg Am. 2002 Mar;27(2):205-15. doi: 10.1053/jhsu.2002.32081. PMID 11901379
- [Result] Orbay JL, Badia A, Indriago IR, Infante A, Khouri RK, Gonzalez E, Fernandez DL. The extended flexor carpi radialis approach: a new perspective for the distal radius fracture. Tech Hand Up Extrem Surg. 2001 Dec;5(4):204-11. doi: 10.1097/00130911-200112000-00004. No abstract available. PMID 16520583
- [Result] Wijffels MM, Orbay JL, Indriago I, Ring D. The extended flexor carpi radialis approach for partially healed malaligned fractures of the distal radius. Injury. 2012 Jul;43(7):1204-8. doi: 10.1016/j.injury.2012.04.002. Epub 2012 Apr 27. PMID 22542167
- [Result] Murray WM, Delp SL, Buchanan TS. Variation of muscle moment arms with elbow and forearm position. J Biomech. 1995 May;28(5):513-25. doi: 10.1016/0021-9290(94)00114-j. PMID 7775488
- [Result] Kim JK, Park JS, Shin SJ, Bae H, Kim SY. The effect of brachioradialis release during distal radius fracture fixation on elbow flexion strength and wrist function. J Hand Surg Am. 2014 Nov;39(11):2246-50. doi: 10.1016/j.jhsa.2014.07.043. Epub 2014 Sep 11. PMID 25218141
- [Result] Lalone E, MacDermid J, Grewal R, King G. Patient Reported Pain and Disability Following a Distal Radius Fracture: A Prospective Study. Open Orthop J. 2017 Jul 31;11:589-599. doi: 10.2174/1874325001711010589. eCollection 2017. PMID 28979578
- [Result] Schneiders W, Biewener A, Rammelt S, Rein S, Zwipp H, Amlang M. [Distal radius fracture. Correlation between radiological and functional results]. Unfallchirurg. 2006 Oct;109(10):837-44. doi: 10.1007/s00113-006-1156-8. German. PMID 16969651
- [Result] Jebsen RH, Taylor N, Trieschmann RB, Trotter MJ, Howard LA. An objective and standardized test of hand function. Arch Phys Med Rehabil. 1969 Jun;50(6):311-9. No abstract available. PMID 5788487
- [Result] Oliveira LC, Pires-Oliveira DA, Abucarub AC, Oliveira LS, Oliveira RG. Pilates increases isokinetic muscular strength of the elbow flexor and extensor muscles of older women: A randomized controlled clinical trial. J Bodyw Mov Ther. 2017 Jan;21(1):2-10. doi: 10.1016/j.jbmt.2016.03.002. Epub 2016 Mar 10. PMID 28167180
- [Result] Ellenbecker TS, Roetert EP, Riewald S. Isokinetic profile of wrist and forearm strength in elite female junior tennis players. Br J Sports Med. 2006 May;40(5):411-4. doi: 10.1136/bjsm.2005.023358. PMID 16632571
- [Result] Seven B, Cobanoglu G, Oskay D, Atalay-Guzel N. Test-Retest Reliability of Isokinetic Wrist Strength and Proprioception Measurements. J Sport Rehabil. 2019 Sep 1;28(7):jsr.2018-0341. doi: 10.1123/jsr.2018-0341. PMID 30676238